CLINICAL TRIAL: NCT04778488
Title: Messung Der Cerebralen Sauerstoffsättigung Mitttels Near-Infrared Spectooxymetrie in Der Reanimation Und Postreanimationsbehandlung
Brief Title: Vienna Near-Infrared Spectroscopy in Cardiac Arrest Study (VINIRSCA)
Acronym: VINIRSCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Emergency Medical Service of Vienna (Unknown)
Responsible Party: Principal Investigator, Sebastian Schnaubelt, MD, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MUV_VINIRSCA
Record Dates: First submitted 2021-02-23; First posted 2021-03-03 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Arrest
Keywords: NIRS; cardiac arrest
MeSH Terms: conditions — Heart Arrest | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Intervention Model Description: Observational cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NIRS diagnostics (Other): NIRS measurement
  Interventions: Device: Near-Infrared-Spectroscopy (NIRS)

INTERVENTIONS:
Device: Near-Infrared-Spectroscopy (NIRS) — Placement of 2 NIRS optodes on the patients' forehead, measurement of NIRS during cardiac arrest and up to 72h post return of spontaneous circulation

SUMMARY:
Measurement of Near-Infrared Spectroscopy (NIRS) during and after out-of-hospital cardiac arrest (OHCA) in the city of Vienna and the tertiary university hospital of the Medical University of Vienna, Austria.

NIRS will be evaluated as a tool for resuscitation quality assessment as well as a prognosticator for cardiac arrest outcomes. Already-existing literature will be taken into account, and already-existing cutoffs and prognosticating values will be assessed and - if eligible - validated in a real-life setting.

DETAILED DESCRIPTION:
Patients suffering from out-of-hospital cardiac arrest (OHCA) and receiving cardiopulmonary resuscitation (CPR) in terms of advanced life support (ALS) in the city of Vienna, Austria, will be included. A special study team will be dispatched to the event sites by the ambulance service. Trained study fellows will include patients by placing NIRS optodes on the patients' forehead as soon as possible during and/or after CPR. Measurements will continue until 72h post return of spontaneous circulation (ROSC) or the patient's death.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* out-of-hospital cardiac arrest

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
near-infrared-spectroscopy | minute 0
  rSO2

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Data can be shared upon reasonable request after assessing and analysing.

REFERENCES:
- [Background] Schnaubelt S, Sulzgruber P, Menger J, Skhirtladze-Dworschak K, Sterz F, Dworschak M. Regional cerebral oxygen saturation during cardiopulmonary resuscitation as a predictor of return of spontaneous circulation and favourable neurological outcome - A review of the current literature. Resuscitation. 2018 Apr;125:39-47. doi: 10.1016/j.resuscitation.2018.01.028. Epub 2018 Feb 2. PMID 29410191
- [Background] Schnaubelt S, Uray T. The need for comprehensive NIRS-measurement from on-scene treatment to post-ROSC phase. Resuscitation. 2019 Nov;144:191-192. doi: 10.1016/j.resuscitation.2019.07.038. Epub 2019 Sep 9. No abstract available. PMID 31513863